CLINICAL TRIAL: NCT00084162
Title: Neurocardiac Control in Major Depression
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040136; 04-M-0136
Record Dates: First submitted 2004-06-08; First posted 2004-06-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-03-17

CONDITIONS: Depression, Involutional
Keywords: PET; Heart Rate Variability; N-Back Task; Isometric Handgrip; MRI; Depression; MDD; Heart
MeSH Terms: conditions — Depressive Disorder, Major; Depression

SUMMARY:
This study will examine how depression may influence the way the brain regulates heart function. Some researchers believe that depression may be a risk factor for some forms of heart disease.

Right-handed healthy volunteers and patients with major depressive disorder who are between 18 and 50 years of age may be eligible for this study. Female candidates must be premenopausal. Patients must currently be experiencing a major depressive episode. All candidates are screened with a medical history and physical examination, electrocardiogram, and blood and urine tests. They are interviewed about their psychiatric and medical history, current emotional state and sleep pattern, and family history of psychiatric disorders. They complete symptoms ratings scales for depression, anxiety, and negative thinking; history of alcohol and tobacco use; level of physical activity; socioeconomic status; overall level of functioning; and, for depressed patients, their depression type. Women candidates have their menstrual phase determined by the timing of their recent menstrual cycles and may undergo testing to determine the time of their ovulation.

Participants undergo the following tests and procedures:

* 12-minute walk/run test - This test measures the subject's general level of cardiorespiratory fitness. In a gymnasium in the NIH Clinical Center, the subject walks or runs as far as he or she can in 12 minutes. Blood pressure is measured before and after the exercise test, and heart rate is measured during exercise with a monitor worn around the chest.
* Magnetic resonance imaging (MRI) - A brain MRI scan is done to obtain pictures of the brain anatomy. Electrocardiogram leads are placed on the subject's chest to measure the electrical activity of the heart during the scanning session. The subject lies on a narrow bed in the scanner, which is a narrow metal cylinder about 6 feet long. The scanning session takes up to 90 minutes.
* Positron emission tomography (PET) - PET scanning produces images of the brain's blood flow. The subject is injected with a radiotracer (small amount of drug labeled with a radioactive substance) that is detected by a special camera to trace blood flow. During the scanning session, the subject lies still on a table. EKG leas are placed on the subject's chest to measure the electrical activity of the heart during the scan. A mask with holes for the eyes, ears, and mouth is placed over the subject's face to keep the head f...

DETAILED DESCRIPTION:
The presence of major depression, with or without pre-existing coronary artery disease, predicts increased mortality from myocardial infarction (MI) and sudden cardiac death (SCD). Decreased parasympathetic vagal outflow, especially in the presence of elevated cardiac sympathetic tone, has been proposed as a mechanism for the increased risk of SCD. Multiple lines of evidence suggests that fronto-limbic areas are actively engaged in the robust optimization of autonomic balance between sympathetic and parasympathetic cardiac outflow over a broad range of cognitive and physical demands. We propose that dysfunction of these forebrain neurocardiac networks in MDD mediates maladaptive cardiac autonomic control and the increased risk of cardiovascular mortality. In this model, neurocardiac control networks exhibit a systemic bias toward increased sympathetic relative to parasympathetic outflow. Increased amygdalar activity in MDD will promote this imbalance. Additionally, dysfunction in posterior orbitofrontal cortex (OFC) and ventral anterior cingulated cortex (ACC), areas associated with abnormal histopathological changes in MDD, will lead to reduced capacity for generating adaptive levels of cardioinhibitory, parasympathetic tone. This reduced capacity in depressives will be evidenced by abnormally large withdrawals of parasympathetic outflow, compared to healthy controls, as cognitive or physical demands increase. This dynamic model is potentially consistent with functional neuroimaging and post mortem histopathological findings in MDD and the knowledge gained through testing this protocol may ultimately elucidate how brain dysfunction in MDD mediates significantly increased clinical risk of spontaneous ventricular arrhythmias and sudden cardiac death.

We propose to combine H (2) (15) O positron emission tomography (PET) and analysis of heart rate variability (HRV) in order to study in vivo the neural structures underlying normal forebrain control of cardiac autonomic function. We further aim to show whether regional functional abnormalities in amygdala, ventral anterior cingulate cortex, and orbitofrontal cortex-areas in which functional abnormalities have been identified in previous neuroimaging studies of major depressives-are associated with impaired modulation of cardiac autonomic function during major depression.

ELIGIBILITY:
* INCLUSION CRITERIA:

Two groups of right-handed subjects, male or premenopausal female, who are drug-naive or who have not received psychotropic drugs for at least 3 weeks (8 weeks for fluoxetine), will be recruited for studies under this protocol: unipolar depressives and healthy controls individually matched to depressives by age, gender and smoking status. Because effective treatment will not be discontinued for the purposes of this protocol, subjects in the patient groups will be identified who have never been treated for or who have discontinued medication due to lack of efficacy, noncompliance, physician order or other reason prior to study entry.

The presence of inclusion and exclusion criteria will be established using both an unstructured clinical interview with a psychiatrist and the Structure Clinical Interview for DSM-IV (SCID). Family history of mental illness will be obtained using the Family Interview of Genetic Studies.

EXCLUSION CRITERIA:

Subjects will be excluded if they have:

serious suicidal ideation or behavior;

inability to provide informed consent;

medical or neurological illnesses likely to affect physiology or anatomy;

a history of drug or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM-IV criteria);

current or past history of other axis I disorders that preceded the onset of MDD;

current pregnancy (documented by pregnancy testing prior to scanning);

current breast feeding;

general MRI exclusion criteria;

vision and/or hearing problems severe enough to interfere with testing.

Exposure within two weeks to medications likely to affect cerebral blood glow or heart rate.

Any condition that may prevent the subject from performing the run/walk test, or

Irregular menstrual cycles so that menstrual phase cannot be reliably determined, or

Any ECG finding that would contraindicate PET scanning or run/walk testing (e.g. non-sinus rhythm, significant tachycardia, ST segment elevation or depression, Q waves) or arrhythmia that would obviate accurate calculation of HRV indices. Cardiology consultation will be obtained for abnormal ECG findings unless it is unequivocally clear in the judgment of the study physician that such consultation is medically unnecessary.

Subjects who are beyond age 50 who are either postmenopausal or perimenopausal are excluded to reduce the biological heterogeneity in autonomic function which may be associated with difference in menstrual status.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2004-03-30; Study Completion 2010-03-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rozanski A, Blumenthal JA, Kaplan J. Impact of psychological factors on the pathogenesis of cardiovascular disease and implications for therapy. Circulation. 1999 Apr 27;99(16):2192-217. doi: 10.1161/01.cir.99.16.2192. PMID 10217662
- [Background] Billman GE. Left ventricular dysfunction and altered autonomic activity: a possible link to sudden cardiac death. Med Hypotheses. 1986 May;20(1):65-77. doi: 10.1016/0306-9877(86)90087-3. PMID 3636581
- [Background] Hull SS Jr, Evans AR, Vanoli E, Adamson PB, Stramba-Badiale M, Albert DE, Foreman RD, Schwartz PJ. Heart rate variability before and after myocardial infarction in conscious dogs at high and low risk of sudden death. J Am Coll Cardiol. 1990 Oct;16(4):978-85. doi: 10.1016/s0735-1097(10)80351-1. PMID 2212380